CLINICAL TRIAL: NCT01846078
Title: Accuracy of Holladay 2 Formula Using IOLMaster Parameters in the Absence of Lens Thickness
Brief Title: Accuracy of Holladay 2 Formula in the Absence of Lens Thickness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Sabong Srivannaboon, Professor Sabong Srivannaboon, Mahidol University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Si343/2012
Record Dates: First submitted 2013-04-30; First posted 2013-05-03 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-04

CONDITIONS: Cataracts
MeSH Terms: conditions — Cataract

ARMS (1):
- Mean absolute errors, median absolute errors (Experimental)
  Interventions: Device: optical biometric measurement (IOLMaster)

INTERVENTIONS:
Device: optical biometric measurement (IOLMaster) — IOLMaster version 5.4 was used to measure the patients' optical biometry by non contact technique.

SUMMARY:
Hypothesis: Holladay 2 formula is still accurate even used without lens thickness data.

ELIGIBILITY:
Inclusion Criteria:

* patients with cataract

Exclusion Criteria:

* previous ocular diseases
* previous ocular surgery

Ages: 44 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2012-06; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
mean absolute error of Holladay2 formula | 6 months
  IOLMaster version 5.4 was used to measure the patients' optical biometry by non contact technique.

CONTACTS AND LOCATIONS:
Locations (1):
- Siriraj Hospital, Bangkok, Thailand

REFERENCES:
- [Background] Narvaez J, Zimmerman G, Stulting RD, Chang DH. Accuracy of intraocular lens power prediction using the Hoffer Q, Holladay 1, Holladay 2, and SRK/T formulas. J Cataract Refract Surg. 2006 Dec;32(12):2050-3. doi: 10.1016/j.jcrs.2006.09.009. PMID 17137982